CLINICAL TRIAL: NCT07248267
Title: Effects of Vojta Therapy on Functional Mobility and Gait Parameter in Children With Down Syndrome
Brief Title: Effects of Vojta Therapy on Functional Mobility and Gait Parameters in Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/AYESHA
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome
Keywords: Downs syndrome, Vojta therapy,Rehabilitation
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial (RCT) designed to compare the effectiveness of vojta therapy on functional mobility and gait parameters on down syndrome children. The study will involve 28 down syndrome children between the ages of 2 and 10. These participants will be randomly divided into two groups. One group will follow Vojta Therapy- Reflexive locomotion that is induced through two positions and 10 stimulus zones. Frequency: 3 times per week for Duration: 30-45 minutes per session. The other group will use Passive range of motion (PROM) and maintain the positioning of child. The control group received conventional physiotherapy which consisted of repetitive sensorimotor exercises
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
  The participant will be blinded throughout the session but the therapist will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator:Vojta Therapy (Experimental): The intervention group received Vojta therapy. Vojta therapy was implemented by stimulating the chest zone, which is located between the 7th and 8th rib, use of additional zones was allowed to support the activation. The starting positions for Vojta therapy were supine or side-lying position with the head turned 30°toward the side being stimulated or side-lying. Patients were treated for 30 min with Vojta therapy and afterwards were mobilized with gait training, if feasible.
  It is recommended that therapy be carried out 30-40 min per day, thrice week. Same types of movements were detected to emerge by applying stimulus to certain points in newborns and s down children
  Vojta defined two main movements:
  Reflex crawling: Stimulating key points on the shoulders and pelvis in this position can help engage the extensor and flexor muscles of the spine, encouraging spinal alignment, limb movement, and balance development.
  Interventions: Other: Vojta Therapy
- repetitive sensorimotor exercises (Placebo Comparator): The intervention should focus on strength training i.e:Core Stability and Trunk Control Exercises:
  Target Muscles: Core stability exercises focus on strengthening the muscles of the trunk, essential for postural control and balance.
  Exercises: Activities like sit-to-stand exercises, balance board training, and core strengthening using resistance bands are commonly used.
  Balance and Coordination Training :Dynamic Balance Exercises: Activities such as standing on one leg, heel-to-toe walking, and using a balance ball help to strengthen lower limb muscles and improve overall coordination.(30) Proprioceptive Activities: Including balance boards and foam pads for standing exercises can enhance proprioceptive feedback, essential for motor planning and gait adjustments
  Interventions: Other: repetitive sensorimotor exercises

INTERVENTIONS:
Other: Vojta Therapy — The intervention group received Vojta therapy. Vojta therapy was implemented by stimulating the chest zone, which is located between the 7th and 8th rib, use of additional zones was allowed to support the activation. The starting positions for Vojta therapy were supine or side-lying position with the head turned 30°toward the side being stimulated or side-lying. Patients were treated for 30 min.Vojta defined two main movements:
  Reflex crawling: Stimulating key points on the shoulders and pelvis in this position can help engage the extensor and flexor muscles of the spine, encouraging spinal alignment, limb movement, and balance development
  Arms: Active Comparator:Vojta Therapy
Other: repetitive sensorimotor exercises — The intervention should focus on strength training i.e:Core Stability and Trunk Control Exercises:
  Target Muscles: Core stability exercises focus on strengthening the muscles of the trunk, essential for postural control and balance.
  Exercises: Activities like sit-to-stand exercises, balance board training, and core strengthening using resistance bands are commonly used.
  Balance and Coordination Training :Dynamic Balance Exercises: Activities such as standing on one leg, heel-to-toe walking, and using a balance ball help to strengthen lower limb muscles and improve overall coordination.(30) Proprioceptive Activities: Including balance boards and foam pads for standing exercises can enhance proprioceptive feedback, essential for motor planning and gait adjustments
  Arms: repetitive sensorimotor exercises

SUMMARY:
This randomized clinical trial investigates the effects of Vojta therapy on functional mobility and gait parameters in children with down syndrome. The study involves 28 male and female children aged 2-10 years old, who will be randomly assigned to one of the two groups i.e. control and experimental group. Key performance outcomes -GMFM 88 and gait outcome assessment -will be assessed both before and after the intervention. The research aims to evaluate the effects of vojta therapy on functional mobility and gait parameters in children with down syndrome. This RCT study will examine the potential key parameters of gait I.e. its spacial parameters that are step length, stride length, stride width, In and out toe and BOS and functional mobility Data will be analyzed through SPSS version 27.00.

DETAILED DESCRIPTION:
This randomized clinical trial provides a detailed effects of Vojta therapy on functional mobility and gait parameters in children with down syndrome. The study is grounded to evaluate the effects of vojta therapy on functional mobility and gait parameters in children with down syndrome. This RCT study will examine the potential key parameters of gait I.e its spacial parameters that are step length , stride length , stride width ,In and out toe and BOS and functional mobility and this study will add potential information in field of pediatrics by examining whether vojta therapy an effective therapeutic intervention over conventional therapeutic plan of care .The study will give the evidence based therapeutic intervention for improvement of DS patient's quality of life and overall mobility .study will be helpful for broader application of reflexive therapies if study will yield supporting results for treating children of down syndrome and their improving their alarming functional mobility and gait commodities.

The study will recruit 28 children with down syndrome between the ages of 2 and 10, who will be randomly assigned to either to control and experimental intervention group for a eight-week period. Performance will be measured using standardized tools that are GMFM 88 and gait outcomes parameters. These assessments will be conducted at baseline before the intervention begins and again immediately following the eight-week intervention given period. The collected data will be analyzed to evaluate the in-between differences of effects of intervention on both groups , with statistical adjustments for baseline values to ensure a robust comparison. The findings are expected to give the evidence based therapeutic intervention for improvement of DS patient's quality of life and overall mobility .study will be helpful for broader application of reflexive therapies if study will yield supporting results for treating children of down syndrome and their improving their alarming functional mobility and gait commodities. Data will be analyzed through SPSS version 27.00.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-10 years old
* Confirmed diagnosis of Down syndrome by pediatric neurologist.
* Written informed consent obtained from parents or guardians.
* Independent standing and walking abilities assessed by GMFM dimension D and E.
* Functional hearing and vision, and understanding of instructions which were necessary for the measurement procedures
* No other physical therapy or interventions within the past three months

Exclusion Criteria:

* Presence of other significant medical conditions (e.g., severe cardiac issues).
* History of orthopedic surgery or significant musculoskeletal issues affecting mobility.
* Any additional neurological disorders that could confound results.
* Patient with Serious cognitive & behavior issues that would interfere with group participation.
* Participation in other clinical trials during the study period

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
1. GMFM-88 scale | 8 weeks
  1. GMFM-88 scale was primary designed to evaluated change in gross motor function of children with CP. At present, 88 items may be used to assess children with DS. Motor functions are grouped in 5 dimensions in GMFM-88: 1) lying and rolling (17 items), 2) sitting (20 items), 3) crawling and kneeling (14 items), 4) standing (13), 5) walking, running and jumping (24 items) [12, 13]. Referring to the guidelines of GMFM-88 assessment for children with DS, the environment should be as familiar to the children as possible, and arranged in such a way to encourage the performance of activities. children performed many tasks spontaneously.. Each task was measured by observation and scored on a 4-point ordinal scale. Value 0 indicated that a child did not initiate the task, 1 point - performed less than 10% of the task, 2 points - a child partially completed a task (10% to< 100%), 3 points - the child completed the task (100%)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Tanveer, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Hashim, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panchal R, Rizvi MR, Sharma A, Ahmad F, Hasan S, Shaik AR, Seyam MK, Uddin S, Ahamed WM, Iqbal A, Alghadir AH. Comparing the effectiveness of the FIFA 11+ warm-up and conventional warm-up in enhancing cyclist performance and mitigating injury risk. Sci Rep. 2025 Mar 19;15(1):9430. doi: 10.1038/s41598-025-91005-z. PMID 40108222